CLINICAL TRIAL: NCT00902785
Title: A Two-Year Exploratory, Observational, Non-Interventional Multicenter Study To Identify Early Markers Of Choroidal Neovascularization In Fellow Eyes Of Patients With Neovascular AMD In One Eye
Brief Title: A Study Of Early Markers Of Choroidal Neovascularization
Status: Terminated | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Other Study IDs: A9011051
Record Dates: First submitted 2009-05-13; First posted 2009-05-15 (Estimated); Last update posted 2010-11-10 (Estimated); Status verified 2010-11

CONDITIONS: Choroidal Neovascularization (CNV); Age-related Macular Degeneration (AMD); Early Markers
Keywords: exploratory; observational; non-interventional study age-related macular degeneration (AMD) choroidal neovascularization (CNV)
MeSH Terms: conditions — Choroidal Neovascularization; Macular Degeneration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- no drug: no drug
  Interventions: Other: no drug

INTERVENTIONS:
Other: no drug — observational no drug

SUMMARY:
Identify early markers of choroidal neovascularization (CNV) in the fellow eye of a patient with CNV in the other eye due to age-related macular degeneration with the expectation of being able to identify patients in need of intervention.

DETAILED DESCRIPTION:
CNV in one eye and dry AMD in the other

ELIGIBILITY:
Inclusion Criteria:

* Sub-, extra- or juxta-foveal choroidal neovascularization (CNV) or macular scar due to AMD in the non-study eye.
* No CNV or geographic atrophy in the study eye.
* Best corrected visual acuity in the study eye of greater than 20/40 or better than 70 ETDRS letters.
* Sufficiently clear ocular media and adequate pupillary dilatation to permit good quality fundus imaging of the study eye.
* Subjects of either sex, aged 50 years.
* Evidence of a signed and dated informed consent document indicating that the subject (or a legally acceptable representative) has been informed of all pertinent aspects of the trial.
* Willing and able to comply with scheduled visits, laboratory tests, and other trial procedures.

Exclusion Criteria:

* Subjects presenting with any of the following will not be included in the study:
* Evidence of manifest CNV by FA, color photography or ICG angiography in the study eye.
* Any prior treatment for CNV to the study eye (excluding vitamins and AREDS formula).
* Significant media opacities, including cataract, which might interfere with visual acuity assessments, or fundus imaging in the study eye. Subjects should not be entered if there is likelihood that they will require cataract surgery within the following 2 years.
* Presence of other causes of choroidal neovascularization in the fellow eye, including pathologic myopia (spherical equivalent of -8 diopters or more negative, or axial length of 25 mm or more), the ocular histoplasmosis syndrome, angioid streaks, choroidal rupture, and multifocal choroiditis.
* Any progressive eye disease other than AMD (eg, glaucoma, diabetic retinopathy) in the study eye.
* Presence of subretinal hemorrhage, serous or hemorrhagic pigment epithelial detachments, subretinal fibrosis or pigment epithelial tears or rips in the study eye.
* Any medical condition that would interfere with the patient's ability to complete the trial.
* Concurrent enrollment in any other observational or interventional clinical study.
* Any treatment with an ocular or systemic investigational agent in the past 60 days for any medical condition.
* Known serious allergies to the dye used in fluorescein angiography or ICG.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * age-related macular degeneration (AMD)
  * choroidal neovascularization (CNV)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-03; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Identify the sequence of change in the chorioretinal interface during the development of CNV and the progression from dry to neovascular AMD. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- Pfizer Investigational Site, Milan, Italy
- Pfizer Investigational Site, Coimbra, Portugal
- Pfizer Investigational Site, Belfast, United Kingdom

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9011051&StudyName=A%20Study%20Of%20Early%20Markers%20Of%20Choroidal%20Neovascularization